CLINICAL TRIAL: NCT05103982
Title: Testing a New Self-help Intervention for Infertility Related Distress: a Pilot Study
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Regina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-108
Record Dates: First submitted 2021-10-20; First posted 2021-11-02 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Infertility, Female
Keywords: infertility-related distress; depression; anxiety
MeSH Terms: conditions — Infertility, Female; Depression; Anxiety Disorders | interventions — Coping Skills

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Coping with Infertility Program (Experimental): The program consists of brief weekly videos, each addressing a particular psychological technique to be implemented that week. Participants receive the videos by email from the researcher and watch them on their own. Each video also assigns a "homework" exercise for the participant to complete that week.
  Interventions: Behavioral: Coping with Infertility Program

INTERVENTIONS:
Behavioral: Coping with Infertility Program — 6 10-minute videos with assigned homework

SUMMARY:
This pilot study will test the effect of a 6-week self-help program in improving fertility-related quality of life as well as anxious and depressive symptoms, in women with infertility.

DETAILED DESCRIPTION:
Twenty women with infertility living in Saskatchewan will be recruited and will be emailed six weekly 10-minute videos, each providing instructions on a new psychological technique that is aimed at addressing the emotional and interpersonal challenges of infertility. Fertility-related quality of life, depressive symptoms, and anxious symptoms will be measured before and after the program. Outcomes will also be measured weekly for three weeks post-intervention. Feedback about how to improve the program will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Has been trying to get pregnant for 12+ months and has failed OR is currently undergoing fertility treatments due to a diagnosis of infertility
* Lives in Saskatchewan, Canada
* Reports a high level of distress related to infertility, as indicated by a FertiQoL score below 52 or at least mild anxious or depressive symptoms (GAD-7 score of 5 or above or PHQ-9 score of 5 or above)

Exclusion Criteria:

* Has a history of suicide attempts
* Is currently experiencing suicidal ideation
* Reports severe depressive symptoms, as indicated by a PHQ-9 score above 19
* Reports severe anxious symptoms, as indicated by a GAD-7 score above 14

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-04-15 (Estimated)

PRIMARY OUTCOMES:
Fertility Quality of Life tool (Fertiqol) | Pre-to-post change in the month following the intervention (post measures assessed 1, 2, 3, and 4 weeks after receipt of last module)
  Pre-to-post change in quality of life related to a diagnosis of infertility. Scores range from 0-100, with higher scores indicating better quality of life

SECONDARY OUTCOMES:
Generalized Anxiety Disorder-7 (GAD-7) | Pre-to-post change in the month following the intervention (post measures assessed 1, 2, 3, and 4 weeks after receipt of last module)
  Pre-to-post change in anxious symptoms; Scores range from 0-21, with higher scores indicating more severe anxiety
Patient Health Questionnaire-9 (PHQ-9) | Pre-to-post change in the month following the intervention (post measures assessed 1, 2, 3, and 4 weeks after receipt of last module)
  Pre-to-post change in depressive symptoms; Scores range from 0-27, with higher scores indicating more severe depressive symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- University of Regina, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Poulter MML, Balsom AA, Gordon JL. Pilot trial of a new self-directed psychological intervention for infertility-related distress. Pilot Feasibility Stud. 2024 Aug 16;10(1):111. doi: 10.1186/s40814-024-01535-y. PMID 39152484